CLINICAL TRIAL: NCT02957838
Title: Mitochondrial Effects of C18:0 Supplementation in Type 2 Diabetics Versus Healthy Controls
Brief Title: Mitochondrial Effects of C18:0 Supplementation in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Collaborators: German Cancer Research Center (Other)
Responsible Party: Principal Investigator, Daniel Pfaff, Principal Investigator, University Hospital Heidelberg
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: S-675/2015
Record Dates: First submitted 2016-10-24; First posted 2016-11-08 (Estimated); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Alteration of Mitochondrial Membrane; Type2 Diabetes; Fatty Acid Deficiency
Keywords: Transferrin Receptor; Type 2 Diabetes; Stearic Acid (C18:0); Mitochondrial Morphology; Crossover Study
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — stearic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-diabetics (Experimental): Non-diabetic volunteers with HbA1c < 6.5%. Subjects will be treated with C18:0 supplementation or mock.
  Interventions: Dietary Supplement: C18:0; Dietary Supplement: mock
- Type 2 Diabetics (Experimental): Type 2 Diabetes according to common definitions, but we exclude insulin-treated Type 2 diabetics because nutritional intervention is more difficult/risky. Subjects will be treated with C18:0 supplementation or mock.
  Interventions: Dietary Supplement: C18:0; Dietary Supplement: mock

INTERVENTIONS:
Dietary Supplement: C18:0 — Receives 24g of C18:0 in a low-fat banana milkshake.
  Other Names: stearic acid; stearic acid, Sigma-Aldrich, product number W303518
Dietary Supplement: mock — Low fat banana milkshake without C18:0 supplement.

SUMMARY:
The purpose of this crossover study is to determine whether nutritional supplementation of C18:0 in humans has mitochondrial effects as shown in Drosophila and human cell culture. We will compare a study cohort of patients with diagnosed type 2 diabetes with non-diabetics. Participants will undergo a 2-day low-fat vegan diet and will then be supplemented with a bolus of C18:0. Changes in the mitochondrial morphology and function of white blood cells will be scored by immunofluorescence and FACS analysis.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether nutritional supplementation of C18:0 in humans has mitochondrial effects as shown in Drosophila and human cell culture. We will compare a study cohort of patients with diagnosed type 2 diabetes with non-diabetics. Participants will undergo a 2-day low-fat vegan diet to reach baseline levels of C18:0 and will then be fed a milkshake supplemented with 24g of C18:0, which corresponds roughly to the C18:0 content of a fast-food meal. Blood samples will be taken at baseline and several hours after intake. We will look at changes in mitochondrial morphology of neutrophils by immunofluorescence, and score mitochondrial function via FACS analysis. Since this study is designed as a crossover study, participants will also receive a mock milk shake after another 2 days of low-fat vegan diet.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes, either dietary treatment or oral medication
* must be able to give consent

Exclusion Criteria:

* insulin treated diabetes mellitus
* severe diseases inducing wasting (e.g. cancer, liver cirrhosis, renal failure)
* conditions of malnourishment
* severe anemia
* pregnancy
* alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-11; Primary Completion 2017-10-06 (Actual); Study Completion 2017-11-18 (Actual)

PRIMARY OUTCOMES:
Changes in Mitochondrial Morphology | 2 days before supplementation, on the day of supplementation at 0, 3 and 6 h
  Mitochondria of neutrophils are stained and scored via immunofluorescence microcsopy, either as "fragmented", "intermediate" or "fused". Statistical calculations will be performed on changes in fragmentation status after treatment.
Changes in Mitochondrial Function | on the day of supplementation at 0, 3 and 6 h
  Mitochondrial membrane potential and ROS production in neutrophils will be analyzed via FACS. Statistical calculations will be performed on changes in the respective levels after treatment.

SECONDARY OUTCOMES:
plasma iron, transferrin, ferritin, ferroportin and hepcidin levels | 2 days before supplementation, on the day of supplementation at 0, 3 and 6 h
  Measurement of iron, transferrin, ferritin, hepcidin and ferroportin from serum at all timepoints via ELISA. Changes in plasma levels will be correlated to primary endpoints.
plasma methylglyoxal levels | 2 days before supplementation, on the day of supplementation at 0, 3 and 6 h
  Methylglyoxal levels in plasma analyzed via liquid chromatography-mass spectrometry. Changes will be correlated to primary endpoints.
plasma fatty acid levels | 2 days before supplementation, on the day of supplementation at 0, 3 and 6 h
  Fatty acids along with other lipid parameters like triglycerides and cholesterol for normalization purposes will be measured.
insulin resistance | 2 days before supplementation, on the day of supplementation at 0, 3 and 6 h
  Insulin and glucose levels will be measured at each time point, HOMA index will be calculated.
diabetic late complications | 2 days before supplementation
  Patients with confirmed HbA1c > 6,5% will be considered diabetic. Then albumin in urine will be measured and diabetic neuropathy will be assessed clinically via NDS/NSS scoring.

CONTACTS AND LOCATIONS:
Overall Officials: Peter P Nawroth, MD, Study Director — University Hospital Heidelberg
Locations (1):
- University of Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
All relevant, collected data will be published.

REFERENCES:
- [Background] Senyilmaz D, Virtue S, Xu X, Tan CY, Griffin JL, Miller AK, Vidal-Puig A, Teleman AA. Regulation of mitochondrial morphology and function by stearoylation of TFR1. Nature. 2015 Sep 3;525(7567):124-8. doi: 10.1038/nature14601. Epub 2015 Jul 27. PMID 26214738